CLINICAL TRIAL: NCT06734182
Title: A Prospective, Single-arm, Multicenter, Phase II Clinical Study on Envafolimab Combined With Disitamab Vedotin And Carboplatin for Resectable, Stage II-III, HER2-Mutant Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant Envafolimab Plus Disitamab Vedotin and Carboplatin in Resectable HER2-Mutant Non-Small-Cell Lung Cancer
Acronym: neovision
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-NSCLC-013
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage II-IIIB; HER2-Mutant; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: single group assignment
Masking Description: No Masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Treatment (Experimental): Patients were treated with subcutaneous Envafolimab injections (300mg, d1, Q3W) combined with intravenous Disitamab Vedotin (2.5mg/kg, d1, Q3W) and carboplatin (AUC5, d1, Q3W)
  Participants receive totally 4 cycles of Envafolimab combined with Disitamab Vedotin and carboplatin during perioperative period
  Interventions: Drug: Envafolimab injections+intravenous Disitamab Vedotin+carboplatin

INTERVENTIONS:
Drug: Envafolimab injections+intravenous Disitamab Vedotin+carboplatin — Biological: Envafolimab 300 mg by subcutaneous injections every 3 weeks (Q3W), given on cycle day 1; Biological: Disitamab Vedotin 2.5mg/kg by IV infusion Q3W, given on cycle day 1;Drug: Corboplatin AUC 5 by IV infusion Q3W, given on cycle day 1;

SUMMARY:
This is a prospective, single-arm, multi-center, phase II clinical study to evaluate the efficacy and safety of Envafolimab injection (PD-L1) combined with Disitamab Vedotin (HER2 ADC) and Carboplatin for resectable, HER2-Mutant, stage II-IIIB, NSCLC.

DETAILED DESCRIPTION:
The eligible patients will receive 4 cycles of subcutaneous Envafolimab injections (300mg, d1, Q3W) in combination with intravenous Disitamab Vedotin (2.5mg/kg, d1, Q3W) and carboplatin (AUC5, d1, Q3W), followed by surgical resection 4-6 weeks after the last dose of neoadjuvant therapy. The tumor tissue samples collected from subjects during the study will be submitted to the authorized central laboratory for evaluation of pathological response and translational research. Dynamic blood samples will be collected at baseline, after neoadjuvant treatment and after surgery for tumor-informed minimal residual disease (MRD) testing. After surgery, patients will be provided with or without adjuvant therapy according to MRD results. Patients with postoperative positive MRD result will be provided with adjuvant treatment after multidisciplinary discussion. The primary endpoint of this study is major pathologic response (MPR) rate. All the subjects will be followed up for overall survival, until death, withdrawal of informed consent or end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Having sufficient understanding of this study and being willing to sign the informed consent form (ICF);
2. Aged 18-75 years, male or female;
3. Treatment-naive, histologically confirmed resectable, stage II, IIIA, IIIB (AJCC staging system, version 9) NSCLC; cTNM stage can be confirmed through PET-CT or pathological biopsy; N2 should be confirmed by mediastinoscopy or EBUS.
4. PET-CT or CT plus MRI should be completed before enrollment;
5. HER2 mutations identified by histological specimens;
6. Measurable lesions based on the response evaluation criteria in solid tumors version 1.1 (RECIST v1.1);
7. Tumor tissue specimens and blood sample available for detection of MRD and biomarkers (the tumor tissue specimens must be freshly obtained or archived samples within 3 months prior to enrollment);
8. ECOG score 0-1;
9. No contraindications to immunotherapy;
10. Adequate organ function:
11. Being willing and able to comply with the visits, treatment plan, laboratory examinations and other study procedures scheduled in the study;
12. Pulmonary function being able to withstand the planned surgery evaluated by surgeons;
13. Women of childbearing potential must undergo a serum pregnancy test within 3 days prior to the first dose and the result must be negative. Female patients of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use highly effective contraceptive methods during the study period and within 180 days after the last dose of study drug

Exclusion Criteria:

1. Presence of locally advanced, unresectable or metastatic disease; unresectable includes the unresectable defined in the Chinese expert consensus on the multidisciplinary diagnosis and treatment for stage III non-small cell lung cancer (2019), including partial stage IIIA and IIIB and all the stage IIIC;
2. Participants with known EGFR sensitive mutations or ALK translocation, KRAS sensitive mutations, BRAF V600E, ROS1 fusions, RET fusions, MET exon 14 alterations and MET amplification, NTRK fusions;
3. Previous treatment with systemic antitumor therapy for early NSCLC, including investigational product;
4. History of (non-infectious) pneumonitis/interstitial lung disease requiring steroid treatment, or ongoing pneumonitis/interstitial lung disease requiring steroid treatment;
5. Active tuberculosis;
6. Active infection requiring systemic treatment;
7. Subjects with any known or suspected autoimmune disorder or immunodeficiency, with the following exceptions: hypothyroidism, hormone therapy is not needed, or well controlled at physiological dose; controlled type I diabetes;
8. Uncontrolled active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] in screening period with HBV-DNA detected higher than the upper limit of normal at the clinical laboratory of the study center); (the subjects with HBV-DNA assay <500 IU/mL within 28 days prior to randomization who have received local standard antiviral therapy for at least 14 days and are willing to receive antiviral therapy continuously during the study can be enrolled); active hepatitis C (defined as positive hepatitis C surface antibody [HCsAb] in screening period and positive HCV-RNA);
9. Known human immunodeficiency virus (HIV) infection (known positive HIV antibody);
10. Vaccination of live vaccine within 30 days prior to the first dose. Including but not limited to the following: parotitis, rubella, measles, varicella/ herpes zoster (varicella), yellow fever, Rabies, Bacille Calmette-Guérin (BCG) and typhoid vaccine (inactivated virus vaccine allowed);
11. Previous use of PD-1/PD-L1 agent or the drug acting on another targeted T cell receptor (e.g., CTLA-4, OX-40);
12. Severe allergic reaction to other monoclonal antibodies;
13. Known serious or uncontrolled pre-existing diseases; including but not limited to cardiovascular events with hemodynamic instability, symptomatic cerebrovascular events, and hepatic cirrhosis above Child-Pugh A within 6 months;
14. Other malignant tumors within 5 years prior to the first dose, except non-small cell lung cancer. The malignant tumors with negligible risk of metastasis or death (e.g., expected disease-free survival > 5 years) and expected to achieve radical outcomes after treatment (e.g., sufficiently treated carcinoma in situ of cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated for radical surgery) can be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2027-06-22 (Estimated); Study Completion 2028-06-22 (Estimated)

PRIMARY OUTCOMES:
MPR rate | up to 7 weeks after neoadjuvant
  Major Pathological Response (MPR) Rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy.

SECONDARY OUTCOMES:
pCR rate | pCR:up to 7 weeks after neoadjuvant;
  Pathological Complete Response (pCR) Rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
ORR | ORR:up to 7 weeks after neoadjuvant;
  Objective Response Rate (ORR) is defined as the percentage of participants achieving complete response (CR) and partial response (PR) for tumor volume reduction and maintaining the minimum duration requirement based on RECIST v1.1
EFS | EFS up to 3 years
  Event Free Survival (EFS) is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.
OS | OS up to 3 years
  Overall survival (OS) is defined as the time from randomization until death from any cause.
Safety evaluation of subjects | Safety: 90 days after the last administration
  Safety: adverse event (AE), abnormal laboratory examination, serious adverse event (SAE) related with the study drug judged using NCI-CTCAE V5.0; surgical feasibility: percentage of procedure delay or cancellation, change of surgical approach, operation time, Incidence of surgical complications；
Molecular progression of ctDNA based on MRD monitoring | up to 3 years
  Molecular progression of ctDNA, defined as the time at which ctDNA mutations were first detected during postoperative MRD haemodynamic monitoring.

OTHER OUTCOMES:
Exploratory analysis of potential biomarkers related with the outcome | up to 3 years
  Exploratory analysis of potential biomarkers related to the outcome (including PD-L1, HER2 expression in tissue specimen, HER2 mutations, and change of ctDNA in peripheral blood sample)

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, China